CLINICAL TRIAL: NCT06816485
Title: Investigation of the Safety and Performance of a Novel PTV Balloon in Patients Undergoing TAVI for Severe Aortic Stenosis
Brief Title: INFLATE Study: Investigation of the Safety and Performance of a Novel PTV Balloon in Patients Undergoing TAVI for Severe Aortic Stenosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biosensors Europe SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-EU-01
Record Dates: First submitted 2025-01-23; First posted 2025-02-10 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Aortic Diseases
Keywords: PTV Balloon; TAVI; Aortic Valve Stenosis; Balloon Aortic Valvuloplasty
MeSH Terms: conditions — Aortic Diseases; Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Single arm, prospective, multi-center, trial designed to enroll approximately 78 patients. All patients will undergo pre-dilatation using at least one study device. Some patients may also undergo post-dilatation with the study device as clinically indicated. All patients will be followed until discharge (maximum 7 days) for data collection. Patients will be enrolled in up to 10 investigational centers in Spain.
  The sample size is based on the expected event rate for patients to be treated with a self-expanding valves only.
  In addition, the study will enroll, in a separate cohort, 15 patients that will be treated with balloon-expanding valves. This cohort will be analyzed and treated separately.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biosensors PTV balloon catheter (Experimental): Patients suffering from a severe aortic stenosis and scheduled for a TAVI.
  Interventions: Device: PTV (Percutaneous Transcatheter Valvuloplasty) Balloon

INTERVENTIONS:
Device: PTV (Percutaneous Transcatheter Valvuloplasty) Balloon — Minimally invasive medical procedure used to replace a diseased aortic valve without the need for open-heart surgery. It is commonly used to treat severe aortic stenosis, a condition in which the aortic valve becomes narrowed and restricts blood flow from the heart to the rest of the body.

SUMMARY:
This clinical investigation is being done to evaluate the safety and effectiveness of a new device, a PTV Balloon, that will be used to open up an area in the heart (the valve) before and potentially after placing a new valve in patients requiring a new heart valve.

The main question it aims to answer is:

What percentage of patients develop new heart conduction problems after using the investigational PTV Balloon for pre-dilatation?

Participants will:

1. Undergo a TAVI procedure, where the PTV Balloon will be used for pre-dilatation and may also be used for post-dilatation.
2. Will be followed up until discharge or up to 7 days, whichever happens first.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic severe calcific stenosis of a native aortic valve with an AVA ≤1.0 cm2 (or AVA index ≤0.6 cm2/m2) AND mean aortic pressure gradient ≥ 40mmHg OR maximal transaortic velocity ≥4.0m/s OR Doppler velocity index ≤0.25 on site-reported echocardiography
2. Local multi-disciplinary Heart Team agrees on indication and eligibility for TAVI
3. Age ≥18 years
4. Patient has signed the Patient Informed Consent Form
5. Patient is willing and able to comply with requirements of the study
6. Patients planned for trans-femoral procedure

Exclusion Criteria:

1. Mean aortic annulus diameter as measured by pre-procedural CT or internal diameter of the bioprosthesis is <16 mm or >30 mm
2. Echocardiographic evidence of intracardiac thrombus, mass or vegetation (site-reported)
3. Significant disease of the aorta that would preclude safe advancement of the TAVI system
4. Severe ilio-femoral vessel disease that would preclude safe performance of the TAVI procedure
5. Severe tricuspid regurgitation and/or failing right heart (site-reported)
6. Severe left ventricular dysfunction with ejection fraction (EF) <20% (site-reported)
7. Evidence of active endocarditis or other acute infections
8. Renal failure requiring continuous renal replacement therapy
9. Untreated clinically significant coronary artery disease requiring revascularization
10. Acute MI ≤30 days prior to the index procedure
11. Symptomatic carotid or vertebral artery disease requiring intervention or carotid/vertebral intervention within the preceding 45 days
12. Cerebrovascular accident (CVA) or transient ischemic attack (TIA) ≤6 months or prior CVA with moderate or severe disability (e.g. modified Rankin scale score >2)
13. History of bleeding diathesis or coagulopathy; acute blood dyscrasias as defined: thrombocytopenia (platelets <80,000/µl), acute anemia (hemoglobin <10 g/dl), leukopenia (WBC <3000/ µl)
14. Severe (greater than 3+) mitral insufficiency (site-reported)
15. Known hypersensitivity to contrast media, which cannot be adequately pre-medicated or contraindication to anticoagulant or anti-platelet medication or to nitinol alloy or to bovine tissue
16. Currently participating in another investigational drug or device study
17. Pregnancy or intend to become pregnant during study participation
18. Unicuspid aortic valve
19. Non-calcified aortic stenosis
20. Identified high risk of coronary occlusion due to Sinus of Valsalva anatomy and/or bulky calcified aortic valve leaflets in close proximity to coronary ostia
21. Isolated Aortic Insufficiency
22. Patients with a permanent pacemaker
23. Patients with pre-existing LBBB, RBBB and AV block 2 and 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the rate of new conduction system abnormalities, including 3rd AV block, LBBB, or RBBB, occurring after pre-dilatation using the study device | During TAVI procedure
  The primary endpoint evaluates the incidence of new conduction system abnormalities that emerge after pre-dilatation using a PTV Balloon, the study device. These conduction system abnormalities include:
  * Third-degree atrioventricular (AV) block: A complete disruption of electrical signals between the atria and ventricles, requiring pacemaker placement in most cases.
  * Left bundle branch block (LBBB): A condition where electrical impulses are delayed or blocked in the left bundle branch, potentially leading to desynchrony in ventricular contraction.
  * Right bundle branch block (RBBB): A delay or blockage of electrical signals in the right bundle branch, which can affect the heart's pumping efficiency.

SECONDARY OUTCOMES:
Successful inflation and deflation of the study device during pre-dilatation | Measured during TAVI procedure
  Rate of study devices successfully inflated and deflated
Balloon rupture during pre-dilatation | measured during TAVI procedure
  absolute number and percentages of balloon ruptures during pre-dilatation
Number of pre-dilatations performed | Measured during TAVI procedure
  Total number
Need for post-dilatation and reason (under expansion, PVL, other) | measured during TAVI procedure
  absolute number and percentages of post-dilatation and reason why
Successful inflation and deflation of the balloon during post-dilatation | measured during TAVI procedure
  Rate of study devices successfully inflated and deflated
Number of post-dilatations performed | measured during TAVI procedure
  absolute number and percentages of post-dilatation
Balloon rupture during post-dilatation | measured during TAVI procedure
  absolute number and percentages of balloon ruptures during post-dilatation
Rate of conduction system abnormalities induced by post-dilatation | measured during TAVI procedure
  Evaluates the incidence of new conduction system abnormalities that emerge after post-dilatation using a PTV Balloon, the study device. These conduction system abnormalities include:
  * Third-degree atrioventricular (AV) block: A complete disruption of electrical signals between the atria and ventricles, requiring pacemaker placement in most cases.
  * Left bundle branch block (LBBB): A condition where electrical impulses are delayed or blocked in the left bundle branch, potentially leading to desynchrony in ventricular contraction.
  * Right bundle branch block (RBBB): A delay or blockage of electrical signals in the right bundle branch, which can affect the heart's pumping efficiency.
Degree of aortic regurgitation (para-valvular) post-dilatation | measured during TAVI procedure
  absolute number and percentages of mild, moderate or severe aortic regurgitation
New onset conduction disorders and arrhythmias at any other times during the procedure | measured during TAVI procedure
  absolute number and percentages of new onset conduction disorders and arrhythmias
Annular rupture | measured during TAVI procedure
  absolute number and percentages of annular ruptures
Usability assessment of the device per case | After TAVI procedure
  Absolute number and percentages within each category of the below scale:
  Unsuccessful Poor Average Good Excellent
All-cause mortality | From enrollment until the patient is discharged (max. 7 days)
  absolute number and percentages of deaths
Cardiovascular mortality | From enrollment until the patient is discharged (max. 7 days)
  absolute number and percentages of cardiovascular deaths
Neurological events (All stroke, stroke disability, transient ischemic attack) | From enrollment until the patient is discharged (max. 7 days)
  absolute number and percentages of neurological events
Procedure or valve related hospitalization | From TAVI procedure until the patient is discharged (max. 7 days)
  absolute number and percentages of hospitalizations
Bleeding | From enrollment until the patient is discharged (max. 7 days)
  absolute number and percentages of bleeding events
Major vascular complications | From enrollment until the patient is discharged (max. 7 days)
  absolute number and percentages of major vascular complications
Major cardiac structural complications | From enrollment until the patient is discharged (max. 7 days)
  absolute number and percentages of major cardiac structural complications
Conversion to open surgery | measured during TAVI procedure
  absolute number and percentages of conversions to open surgery
Valve malposition (valve migration, valve embolization, ectopic valve deployment) | measured during TAVI procedure
  Absolute number and percentages of valve malpositions

CONTACTS AND LOCATIONS:
Locations (7):
- Spain (7):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid (HCUV), Valladolid